CLINICAL TRIAL: NCT03146910
Title: Swiss Primary Biliary Cholangitis Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Other Study IDs: SASL39 - Swiss PBC Cohort
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: PBC; Primary Biliary Cholangitis
Keywords: PBC; Primary Biliary Cholangitis; Cohort; AILD
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — 1. Serum (BD Vacutainer® SST II Advance)
  2. RNA (PAXgene™ Blood RNA tube- 762165)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Research project in which biological material is sampled and health-related medical data is collected. In addition, already existing health-related medical data are used for further research. Coded data are used.

DETAILED DESCRIPTION:
Enrolment visit and one follow-up visit at least once a year are planned.

Whole blood is collected for biobanking once a year. Optionally, if available and collected during normal clinical procedures, liver fragments are obtained.

To collect high quality prospective data on a rare disease in order to elucidate epidemiology, natural history, response to treatment and outcome. In addition, the biobank allows addressing specific scientific issues on a variety of open questions. The cohort will provide a platform for carrying out scientific research projects on PBC. In addition, the cohort will allow collaboration with reference networks on PBC abroad.

ELIGIBILITY:
Inclusion Criteria:

* diagnose of Primary biliary cholangitis (according to EASL Clinical Practice Guidelines: management of cholestatic liver diseases).
* Subjects with isolated anti-mitochondrial antibodies and/or isolated PBC-specific anti-nuclear antibodies are also included
* Patients/subjects aged at least 18 years and living in Switzerland are included

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Primary biliary cholangitis according to recognized criteria (European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases). Subjects with isolated anti-mitochondrial antibodies and/or isolated PBC-specific anti-nuclear antibodies are also included. Patients/subjects aged at least 18 years and living in Switzerland are included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease course | 3 years
  Observing disease course
Disease features | 3 years
  Observing disease features in Swiss population and see if they are similar to other countries'
Response to treatment | 3 years
  Observing response to treatment
Overall survival | 3 years
  Observing overall survival
Transplantation-free survival rate | 3 years
  Observing transplantation-free survival rate

CONTACTS AND LOCATIONS:
Locations (13):
- Switzerland (13):
  - Fondazione Epatocentro Ticino, Lugano, Canton Ticino
  - Gastroenterologie und Hepatologie, Clarunis - Universitäres Bauchzentrum Basel, Basel
  - Inselspital, Bern
  - Spital Bülach, Bülach
  - Kantonsspital Graubünden, Chur
  - Hôpitaux Universitaires de Genève, Service de Gastroentérologie & Hépatologie, Département des Spécialités, Geneva
  - CHUV: Centre hospitalier universitaire vaudois, Lausanne
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - EOC Ospedale Regionale di Lugano - Italiano, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No